CLINICAL TRIAL: NCT01318226
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Multicenter, Parallel Group Study to Evaluate the Safety and Analgesic Activity of ATx08-001 When Administered to Subjects With Postherpetic Neuralgia
Brief Title: Study to Evaluate the Safety and Analgesic Activity of ATx08-001 in Subjects With Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aestus Therapeutics (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Symbiance, Inc (Unknown); Parallax Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX-1001; R44NS059140 (NIH)
Record Dates: First submitted 2011-03-10; First posted 2011-03-18 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Postherpetic Neuralgia
Keywords: postherpetic neuralgia; shingles; analgesia; neuropathic pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Agnosia; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo will be administered as a 6mm white film coated tablet, twice a day approximately every 12 hours over an 8 day period. Placebo is identical in appearance to the ATx 08-001 tablet.
  Interventions: Drug: Placebo
- ATx08-001 2.5 mg bid (Experimental): ATx08-001 will be administered as a 6mm white film coated tablet of 2.5 mg strength, to be taken orally at a dose of 2.5 mg, twice a day approximately every 12 hours over an 8 day period.
  Interventions: Drug: ATx08-001
- ATx08-001 7.5 mg bid (Experimental): ATx08-001 will be administered as a 6mm white film coated tablet of 2.5 mg strength, to be taken orally at a dose of 7.5 mg, twice a day approximately every 12 hours over an 8 day period.
  Interventions: Drug: ATx08-001

INTERVENTIONS:
Drug: ATx08-001 — ATx08-001 will be administered as a 6mm white film coated tablet of 2.5 mg strength, to be taken orally at a dose of 2.5 mg or 7.5 mg, twice a day approximately every 12 hours over an 8 day period.
  Arms: ATx08-001 2.5 mg bid; ATx08-001 7.5 mg bid
Drug: Placebo — Placebo will be administered as a 6mm white film coated tablet, twice a day approximately every 12 hours over an 8 day period. Placebo is identical in appearance to the ATx 08-001 tablet.
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, multiple-dose, multicenter, parallel-group study to evaluate the analgesic activity of ATx08-001, a novel selective peroxisome proliferator-activated receptor modulator (SPPARM), in subjects with moderate-to-severe postherpetic neuralgia pain. Eligible subjects will be randomized to receive either placebo or Atx08-001. Study drug will be administered orally twice a day for 7 days. Subjects will be evaluated for neuropathic pain intensity at regular intervals over a 6 hour period on Day 1 following the first dose of study drug. They will then be discharged from the clinic and will complete diary assessments of pain severity twice a day at home. Subjects will be asked to return to the clinic on Day 8 to complete their last set of pain evaluations.

DETAILED DESCRIPTION:
Aestus has identified a novel selective peroxisome proliferator-activated receptor modulator (SPPARM), with promising potential for the treatment of neuropathic pain. PPARs are nuclear receptors that control many cellular and metabolic processes and are readily modulated by a variety of different drugs. Drugs modulating this target have been shown to improve blood glucose levels and levels of blood lipids, and may reduce the risk of atherosclerosis.

The primary objective of the study is to evaluate the safety and analgesic efficacy of ATx08-001 at doses of 2.5 mg bid and 7.5 mg bid compared to placebo for the control of moderate-to-severe postherpetic neuralgia (PHN) pain.

The secondary objectives are:

* To determine the approximate time to onset of analgesia following administration of study drug
* To determine the approximate duration of analgesia following study drug administration
* To determine the percentage of treatment responders among subjects receiving ATx08-001

Subjects will be given a diary and instructed to record their postherpetic neuralgia pain severity on a Numerical Pain Rating Scale (NPRS - 12) "over the past 12 hours" on a 0 - 10 scale with "0" being no pain and "10" being the most severe pain the subject could imagine, each morning and night for three consecutive days prior to returning for the Treatment Visit.

The Treatment Visit will consist of an in-clinic 6-hour observation period. To be eligible for dosing, immediately before dosing subjects must report a baseline score of 4 or greater on the following Numerical Pain Rating Scale (NPRS-NOW) question: "How would you rate your pain RIGHT NOW using a zero to ten scale, where zero equals no pain and ten is the worst pain you can imagine." Qualified subjects will be administered study drug followed by a 6-hour observation in-clinic period. In addition to the Baseline pain intensity assessment conducted just prior to drug administration (Time 0), pain intensity scores (pain right now) will be assessed using the NPRS-NOW at 30 minutes, 1, 2, 3, 4, and 6 hours following study drug administration. Pain relief compared with Baseline will be assessed at those same time points using a 5-point numerical pain relief (NPR) scale, where 0 = no relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, and 4 = complete relief.

Subjects will be discharged from the clinic at the end of the 6-hour observation period and will be instructed to record postherpetic neuralgia pain severity (NPRS-NOW scores) and pain relief (PAR scores) at 8, 10 and 12 hours following dosing in a diary.

ELIGIBILITY:
Inclusion Criteria:

* Is able to provide written informed consent prior to study entry
* Is male or female, 18 - 85 years of age
* Has a diagnosis of postherpetic neuralgia that has been present for at least 3 months since the resolution of the skin rash (shingles), and has been associated with at least moderate pain
* Has a body mass index (BMI) between 17 and 36, inclusive
* Has on average postherpetic neuralgia pain severity of at least "4" on the 11-point NPRS-12 scale over three days prior to the Treatment Visit.
* At the Treatment Visit, entry into the study for dosing will require a baseline score of 4 or greater on the following 'Numerical Pain Rating Scale' (NPRS-NOW): "How would you rate your pain RIGHT NOW using a zero to ten scale, where zero equals no pain and ten is the worst pain you can imagine." If the subject fails to qualify for the Treatment Visit because of a baseline pain score below 4, he or she may return on any day within a fourteen day period to attempt to qualify again. A subject will be allowed a maximum of two reassessments to qualify on the basis of the NPRS-NOW scale.
* Female subjects must be of non childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or must be using adequate contraception (practicing one of the following methods of birth control):
* Total abstinence from sexual intercourse (minimum of one complete menstrual cycle before study entry),
* A partner who is physically unable to impregnate the subject (e.g., vasectomized)
* Contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to study drug administration,
* Intrauterine device (IUD), or
* Double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)
* If female of childbearing potential, subject must have a negative serum pregnancy test at screening
* Able to communicate meaningfully with the study observer and staff
* No known allergies to study medication

Exclusion Criteria:

* Has another source of moderate-to-severe pain apart from the postherpetic neuralgia that might be confused with the PHN pain
* Is actively abusing alcohol or drugs
* Is unable to refrain from alcohol for a period beginning 24 hours prior to the treatment visit until the end of the study
* Is scheduled to undergo any surgical procedures during the period of study duration
* Has a history of any active serious medical conditions including cancer (with the exception of benign uterine dysplasia or removed skin carcinomas), cardiovascular, respiratory, renal, hepatic, gastrointestinal, endocrine, immunologic, hematologic, neurologic or psychiatric disease that would contraindicate study participation
* Has moderate to severe (New York Heart Association [NYHA] Class 3 or 4) heart failure defined as heart failure which significantly limits physical activity by provoking fatigue, palpitations or dyspnea.
* Has a history of either type 1 or type 2 diabetes mellitus
* Has taken a fixed scheduled opioid regimen within 3 days prior to the Treatment Visit. A fixed scheduled regimen of another type of analgesic, e.g., nonsteroidal antiinflammatory drug (NSAID) or an adjuvant analgesic will be allowed as long as the dose and schedule of administration were not changed for at least 2 weeks prior to dosing.
* Has used a short-acting "as needed" opioid less than 12 hours prior to dosing or an "as needed" NSAID dose less than 24 hours prior to dosing
* Has used extended duration oral analgesics up to 48 hours prior to the Treatment Visit
* Has applied lidocaine patches or dermal analgesics within 7 days prior to the Treatment Visit
* Has received an anesthetic block within two weeks of the Screening Visit
* Has received any prior neurolytic nerve block in the area of the PHN pain
* Is taking tricyclic, selective serotonin reuptake inhibitor (SSRI) or serotonin and noradrenaline reuptake inhibitor (SNRI) antidepressants for PHN (or for indications other than pain) and the dosage has been changed within 14 days of the Treatment Visit. Only subjects on stable doses from at least 14 days prior to the Treatment Visit through the duration of the study will be eligible to participate
* Is taking gabapentin (Neurontin), pregabalin (Lyrica), or duloxetine (Cymbalta) and the dosage has been changed within 14 days of the Treatment Visit. Only subjects receiving stable doses for at least 14 days prior to the Treatment Visit and are willing to continue taking the same doses for the duration of the study will be eligible to participate
* Has taken any medication that is a substrate of the cytochrome P450 enzyme CYP2C9 within 4 days of dosing with study drug or is unwilling to refrain from such medications through the course of study drug treatment
* Has taken any prescription or over-the-counter medication within three days prior to the Treatment Visit, or herbal agents or other nutraceutical products within 14 days prior to the Treatment Visit, that in the opinion of the Investigator would be expected to confound the analgesic response
* Has documented liver failure or a serum ALT, AST, alkaline phosphatase, or GGT greater than 2.5 times the upper limit of normal, or total bilirubin greater than 1.5 times the upper limit of normal without a known, not clinically significant explanation
* Has a Brain Natriuretic Peptide (BNP) level > 150 pg/mL
* Has a history of poorly controlled hyperthyroidism or hypothyroidism or Thyroid Stimulating Hormone (TSH) levels that are < 0.3 or > 5.5 µlU/mL
* Has moderate or severe renal failure defined as a calculated creatinine clearance of < 60mL/min from the Cockcroft & Gault formula
* Has a clinically significant abnormality on 12-lead electrocardiogram
* Has a known history of a positive Human Immunodeficiency Virus (HIV) antibody test or known HIV infection
* Has a history of a positive Hepatitis B core antibody, or anti-HCV antibody test
* Has previously been admitted to this study
* Has received an investigational medication within 30 days prior to the Treatment Visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Sum of the Pain Intensity Difference at 6 hours (SPID-6) | Baseline to 6 hours after initial dose
  Pain intensity will be measured with a numerical pain rating scale assessing "pain right now" where 0=no pain and 10=worst pain you can imagine. Pain intensity difference (PID) will be calculated by subtracting the pain intensity score at each time point from the Baseline pain intensity score. The SPID (Sum of the Pain Intensity Difference) score will be calculated by summing weighted PID scores over 6 hours, where the weight assigned to each PID score is equal to the elapsed time (in hours) since the previous scheduled evaluation time point.
12-Hour Pain Intensity Scores Assessed with a Numerical Pain Rating Scale (NPRS-12) | Seven Day Treatment Period
  Pain intensity over the 7 day treatment period will be assessed using a numerical pain rating scale that assesses the subject's perception of average pain intensity over the past 12 hours (NPRS-12). The NPRS-12 will be completed by the subject every morning and evening for seven days. Pain intensity will be measured using an 11-point numerical scale where 0 = no pain and 10 = worst pain imaginable.

SECONDARY OUTCOMES:
Summed Pain Intensity Difference (SPID) at Various Time Points | 1 hour period, 2 hour period, 4 hour period, 8 hour period, 10 hour period, 12 hour period
  Pain intensity is measured with a numerical pain rating scale assessing "pain right now" where 0=no pain and 10=worst pain imaginable. Pain intensity difference (PID) is calculated by subtracting the pain intensity score at each time point from the Baseline pain intensity score. SPID (Sum of the Pain Intensity Difference) score will be calculated by summing weighted PID scores over the time period, where the weight assigned to each PID score is equal to the elapsed time since the previous scheduled time point. SPID will be assessed at 1,2,4,8,10 and 12 hours following first dose.
Total Pain Relief (TOTPAR) at 6 hours | Baseline to 6 hours after initial dose
  Pain relief will be assessed at 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours following study drug administration using a numerical pain relief scale (NPR), where 0 = no relief, 1=little relief, 2=some relief, 3=a lot of relief, and 4 = complete relief. Total Pain Relief (TOTPAR) is calculated by summing the hourly NPR scores using the area under the NPR curve. TOTPAR will be assessed from Baseline to 6 hours following dosing.
Pain Intensity Difference (PID) at Various Time Points | Baseline (prior to first dose), 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours after initial dose
  Pain intensity scores (assessing pain right now) will be recorded using a numerical pain rating scale for pain right now (NPRS-NOW) at 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours following study drug administration. Pain will be rated on an 11-point numerical scale where 0 = no pain and 10 = worst pain imaginable.
Pain Relief (PAR) at Various Time Points | Baseline (prior to first dose), 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours after initial dose
  Pain relief compared with Baseline will be assessed at 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours following study drug administration using a 5-point numerical pain relief (NPR) scale, where 0 = no relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, and 4 = complete relief.
Subject-rated Global Evaluation of Study Medication at 6 hours | 6 hours after initial dose (or immediately prior to receiving rescue medication)
  At 6- hours following the first dose of study medication the subject will be asled to assess their overall impression of the study medication and rate it on a 5-point scale, where 0 = poor, 1 = fair, 2 = good, 3 = very good, 4 = excellent. Subjects will rate the study medication based on their perception of its efficacy and tolerability.
Subject-rated Global Evaluation of Study Medication at the Follow-up Visit on Day 8 | Follow-up Visit
  At the follow-up visit on Day 8, the subject will be asked to assess their overall impression of the study medication and rate it on a 5-point scale, where 0 = poor, 1 = fair, 2 = good, 3 = very good, 4 = excellent. Subjects will rate the study medication based on their perception of its efficacy and tolerability.
Total Pain Relief (TOTPAR) at 12 hours | Baseline to 12 hours
  Pain relief will be assessed at 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours following study drug administration using a numerical pain relief scale (NPR), where 0 = no relief, 1=little relief, 2=some relief, 3=a lot of relief, and 4 = complete relief. Total Pain Relief (TOTPAR) is calculated by summing the hourly NPR scores using the area under the NPR curve. TOTPAR will be assessed until 12 hours after dosing.
Time to First Rescue Medication Use | Baseline to 6 hours after initial dose
  Time to the first rescue medication use will be calculated by determining the number of minutes between the time the first dose of study drug was taken and the time of the first request for rescue analgesia. For subjects who did not take any rescue medication, the time to the first rescue medication use will be censored at the time of the final pain assessment during the observation period. If the time to event is greater than 6 hours, subjects will be assigned a time of 6 hours and will be considered censored in the statistical analysis.
Treatment Responders at 6 Hours | Baseline to 6 hours after initial dose
  Subjects will be considered responders for the 6-hour observation period if they demonstrate at least 30% improvement in NPRS-NOW score, and a Pain Relief score > 1, and a Global Evaluation Score of 2, 3, or 4.
Neuropathic Pain Scale (NPS) Ratings at Various Time Points | Baseline (prior to initial dose), and at 1, 2, 4, and 6 hours and follow up visit
  The Neuropathic Pain Scale (NPS) is an instrument designed to measure 6 different pain qualities (sharp, dull, hot, cold, sensitive, and itchy), the overall intensity of the pain, its subjective unpleasantness and two ratings of special characteristics (deep and surface pain) to characterize most manifestations of neuropathic pain on an 11-point categorical scale. The maximum total score is 100, with higher scores indicating greater severity.
Tactile Allodynia Assessment at Various Time Points | Baseline (prior to initial dose), and at 1, 2, 4, and 6 hours and follow up visit
  Tactile Allodynia measures the patient's perception of innocuous stimuli as painful. A standard paintbrush (supplied by the Sponsor) will be brushed over a 5 cm area of skin at the site of maximum pain sensitivity and the subject will rate the severity of pain on a 100 mm VAS scale. The assessment will be performed on symmetrical dermatomes and compared.
Treatment Responders for the Treatment Period | Baseline to Day 8
  Subjects will be considered responders for the 7-Day Treatment Period if they demonstrate a 30% improvement in NPRS-12 compared to the average NPRS-12 score from the three day period before the Treatment Visit, and if they report a Global Evaluation score of 2, 3, or 4.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Radiant Research, Chandler, Arizona
  - Premier Research Center, Peoria, Arizona
  - Homestead Clinical Research, Cutler Bay (Miami), Florida
  - San Marcus Research Clinic, Miami, Florida
  - Boston Clinical Trials, Boston, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Radiant Research, Las Vegas, Nevada
  - Radiant Research, Dallas, Texas